CLINICAL TRIAL: NCT00014131
Title: Vaccine Biotherapy Of Cancer: Autologous Tumor Cells And Dendritic Cells As Active Specific Immunotherapy In Patients With Stage IV Renal Cell Carcinoma
Brief Title: Vaccine Therapy in Treating Patients With Kidney Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: change in corporate priorities
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068493; HOAG-VACCINE-RN (Other: Hoag Cancer Center at Hoag Memorial Hospital Presbyterian); NCI-V01-1647 (Other: National Cancer Institute)
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological/Vaccine (Experimental): Biological/Vaccine: therapeutic autologous dendritic cells. Apheresis procedure collects peripheral blood mononuclear cells (PBMC) for the production of dendritic cell, which are admixed with irradiated tumor cells from autologous tumor cell line for vaccine product.
  Interventions: Biological: Biological/Vaccine: therapeutic autologous dendritic cells.

INTERVENTIONS:
Biological: Biological/Vaccine: therapeutic autologous dendritic cells. — Biological/Vaccine: therapeutic autologous dendritic cells. Apheresis procedure collects peripheral blood mononuclear cells (PBMC) for the production of dendritic cell, which are admixed with irradiated tumor cells from autologous tumor cell line for vaccine product.

SUMMARY:
RATIONALE: Vaccines made from a patient's white blood cells and tumor cells may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy in treating patients who have recurrent or stage III or stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of immunization with in vitro-treated autologous tumor cells and dendritic cells with sargramostim (GM-CSF) in patients with stage III or IV or recurrent renal cell cancer.
* Determine the frequency of conversion of delayed tumor hypersensitivity tests in these patients treated with this regimen.
* Determine the progression-free and overall survival of these patients treated with this regimen.
* Determine the objective tumor response rate in patients who still have measurable disease at the time they are treated with this regimen.

OUTLINE: Patients are stratified according to measurable disease at the time vaccine therapy is initiated (yes vs no).

Patients undergo tumor cell harvest. Patients with multiple persistent sites of metastatic disease following harvest receive systemic therapy (biologic therapy and/or chemotherapy) during tumor cell line expansion. Over 2-4 months, the tumor cell line is expanded, treated with interferon gamma, and irradiated.

Patients undergo leukapheresis to obtain peripheral blood mononuclear cells (PBMC). The PBMC are incubated over 7 days with sargramostim (GM-CSF) and interleukin-4 to produce dendritic cells (DC). The DC are incubated over 2-3 days with the irradiated tumor cells from the autologous tumor cell line for antigen loading of the DC.

Patients undergo delayed tumor hypersensitivity testing 1 week prior to vaccination and again at week 4. Patients receive vaccine therapy comprising autologous treated tumor cells and DC suspended in GM-CSF subcutaneously weekly for 3 weeks. Vaccine therapy continues monthly for 5 months in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year and then every 3 months for 4 years.

PROJECTED ACCRUAL: A total of 80 patients (40 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Stage III or IV disease involving invasions beyond Gerota's fascia, regional lymph node involvement, or distant metastases OR
  * Recurrent disease involving lymph node metastases or soft tissue nodules
* Measurable disease by anatomic-based radiological tests (unless no evidence of disease as documented by prior surgery)
* Planned resection of tumor to establish an autologous tumor cell line
* No active CNS metastases such as brain metastases, spinal cord compression, or leptomeningeal disease

  * Prior brain metastases or spinal cord compression allowed provided there is radiographic evidence of lack of progression and no requirement for pharmacologic doses of corticosteroids

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 4 months

Hematopoietic:

* Hematocrit greater than 25%
* Platelet count greater than 100,000/mm3
* No ongoing transfusion requirements
* No active blood clotting or bleeding diathesis

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* Albumin at least 3.0 g/dL
* No significant hepatic dysfunction

Renal:

* Creatinine no greater than 2.0 mg/dL
* No significant renal dysfunction

Cardiovascular:

* No underlying cardiac disease associated with New York Heart Association class III or IV heart function
* No unstable angina related to atherosclerotic cardiovascular disease

Other:

* No other malignancy within the past 5 years except carcinoma in situ, basal cell or localized squamous cell skin cancer, or localized prostate cancer
* No active infection
* No other active medical condition that could be eminently life threatening
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Other prior putative vaccines allowed
* Recovered from prior biologic therapy
* No concurrent biologic therapy except epoetin alfa for patients with hematocrit less than 36%

Chemotherapy:

* At least 3 weeks since prior chemotherapy and recovered
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No concurrent corticosteroids

Radiotherapy:

* At least 3 weeks since prior radiotherapy (including whole-brain radiotherapy) and recovered
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* Concurrent bisphosphonates allowed for patients with lytic bone metastases
* No concurrent digoxin or other medications designed to improve cardiac output
* No other concurrent anticancer therapy or investigational therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2001-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Conversion of the delayed-type hypersensitivity (DTH) skin test as measured by metric skin ruler at week 4 and month 6 during vaccine therapy | week 4 and month 6 during vaccine therapy
Tumor response (partial response or complete response) as measured by RECIST at months 2 or 3 and 6 during study treatment, and 6 months after study completion | months 2 or 3 and 6 during study treatment, and 6 months after study completion
Progression-free survival as measured by RECIST at months 2 or 3 and 6 during study treatment and every 6 months after study completion | months 2 or 3 and 6 during study treatment and every 6 months after study completion
Event-free survival as measured by RECIST at months 2 or 3 and 6 during study treatment and every 6 months after study completion | months 2 or 3 and 6 during study treatment and every 6 months after study completion
Overall survival beginning at the date of study entry | 5 years or until death, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Cancer Center at Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States